CLINICAL TRIAL: NCT03226613
Title: Advancing New Modalities for the Detection of Oropharyngeal Cancer: Transcervical Ultrasound and HPV16 E6 Antibodies
Brief Title: New Modalities for Detection of Oropharyngeal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Krystle Kuhs, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 170297
Record Dates: First submitted 2017-07-13; First posted 2017-07-24 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Human Papillomavirus Positive Oropharyngeal Squamous Cell Carcinoma; Oropharynx Cancer; Base of Tongue Carcinoma; Tonsil Cancer
Keywords: Human Papillomavirus; Oropharyngeal Cancer; Base of Tongue Cancer; Tonsil Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Tonsillar Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Masking Description: Investigators conducting the ultrasound study will be masked as to the characteristics/location of patient's tumor in order to determine feasibility of identifying oropharyngeal cancers as a sole imaging technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with suspected or known oropharyngeal cancer (Experimental): Patients with either known or suspected oropharyngeal cancer will be asked to undergo a transcervical ultrasound and to provide a blood and oral rinse specimen.
  Interventions: Procedure: Transcervical Oropharyngeal Ultrasound; Procedure: Oral Rinse Collection; Procedure: Blood Draw

INTERVENTIONS:
Procedure: Transcervical Oropharyngeal Ultrasound — One time approximately 15 minute ultrasound will be conducted at the time of clinic visit, focusing on the base of tongue and palatine tonsil via transcervical approach.
  Other Names: Phillips Lumify System (L12-4 transducer)
Procedure: Oral Rinse Collection — Patients will provide a one time oral rinse specimen using a non-alcoholic mouthwash at the time of clinic visit. The participant will be instructed to swish vigorously for 5 seconds and then gargle 5 seconds. The participant will be asked to repeated the swish and gargle (5 seconds each) three times for a total of 30 seconds and then expel the wash in a 10mL conical tube.
Procedure: Blood Draw — A certified phlebotomist will perform a one time blood draw of 10mL at the time of clinic visit from each participant for purposes of HPV serologic testing.

SUMMARY:
Background: The incidence of human papilloma virus-driven oropharyngeal cancer (HPV-OPC), a type of head and neck cancer, is rapidly increasing within the US. Currently, there are no screening methods for early detection. HPV16 E6 antibodies combined with ultrasound imaging may be a promising method for early detection of HPV-OPC. However, prior to testing HPV16 E6 antibodies and ultrasound for HPV-OPC screening, larger studies are needed to further validate the utility of these methods in the diagnostic setting among patients with suspected and/or symptomatic HPV-OPC.

Objective/Hypothesis: To investigate two promising screening modalities for the detection of HPV-OPC, transcervical ultrasound and HPV16 E6 antibodies. The investigators hypothesize that both ultrasound and HPV16 E6 antibodies will be highly sensitive for the detection of symptomatic HPV-OPC.

Specific Aims: (1) Determine the sensitivity of ultrasound to characterize OPC tumors compared to current standard imaging modalities among patients with suspected or confirmed OPC. (2) To determine the sensitivity and specificity of HPV16 E6 antibodies for HPV-OPC. (3) Determine the sensitivity of ultrasound to detect HPV-OPC compared to current standard imaging modalities among patients that present with a neck mass and unknown primary tumor.

DETAILED DESCRIPTION:
50 patients with suspected or confirmed OPC will undergo a transcervical ultrasound during their first visit at the Vanderbilt Head and Neck Clinic in addition to other imaging modalities (CT, MRI and/or PET) as indicated as part of routine clinical care; patients will also be asked to provide a blood specimen. Ultrasound exams will be performed by a clinician blinded to details of the case. All patients will have a CT as part of their diagnostic work-up. Sensitivity of ultrasound to detect tumors identified by CT will be determined. Approximately 40% of patients are expected to test negative on CT requiring MRI and/or PET imaging. Among this subset, the sensitivity of ultrasound to detect tumors identified by either PET and/or MRI will be determined. Tumor size will be determined by 3 ultrasound measurements along the largest diameter of the tumor; agreement between ultrasound and the clinical imaging modalities will be calculated. The investigators will recruit an additional 78 OPC patients with pre-treatment serum banked within the Vanderbilt Head and Neck Cancer Biorepository (18 HPV-negative, 60 HPV-OPC) for HPV serologic analyses; total: 128 samples. Sensitivity and specificity of HPV16 E6 antibodies for detecting HPV-OPC will be calculated. As an exploratory aim, the proportion of tumors undetectable by CT, PET, and MRI, but detected by ultrasound will be determined.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Suspected or confirmed oropharyngeal cancer
* Previously untreated cancer
* First cancer diagnosis

Exclusion Criteria:

* No to any of the inclusion criteria
* Under 21 years of age
* Inability to provide blood or oral rinse specimen

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Detection of tumor via transcervical ultrasound | 1 day at time of clinic visit
  Ability to detect oropharyngeal tumor via ultrasound will be a primary outcome of the study. Characteristics including ability to detect tumor, tumor size, and tumor location will be recorded at time of ultrasound. The ultrasound findings will then be compared to other imaging modalities used as standard work-up (CT/MRI). This comparison will be used to determine sensitivity of ultrasound for detection of oropharyngeal tumors.

SECONDARY OUTCOMES:
HPV Serology | Through study completion, an average of 1 year
  Both serum samples and oral rinse specimens will be shipped to German Cancer Research Center, Heidelberg (DKFZ) for blinded analysis of HPV antibodies. The samples will be completely de-identified prior to shipment and thus, there will be no way for the testing laboratory to link the specimens back to the patients. A random sample of blinded duplicates (10%) will be included as part of quality control. Seroreactivity against the HPV16 E6 protein will be determined using multiplex serology, an antibody detection method based on a glutathione S-transferase capture ELISA in combination with fluorescent bead technology.

CONTACTS AND LOCATIONS:
Overall Officials: Krystle A Kuhs, PhD, Principal Investigator — Assistant Professor for Division of Epidemiology and Department of Otolaryngology, Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaturvedi AK, Engels EA, Pfeiffer RM, Hernandez BY, Xiao W, Kim E, Jiang B, Goodman MT, Sibug-Saber M, Cozen W, Liu L, Lynch CF, Wentzensen N, Jordan RC, Altekruse S, Anderson WF, Rosenberg PS, Gillison ML. Human papillomavirus and rising oropharyngeal cancer incidence in the United States. J Clin Oncol. 2011 Nov 10;29(32):4294-301. doi: 10.1200/JCO.2011.36.4596. Epub 2011 Oct 3. PMID 21969503
- [Background] Coquia SF, Hamper UM, Holman ME, DeJong MR, Subramaniam RM, Aygun N, Fakhry C. Visualization of the Oropharynx With Transcervical Ultrasound. AJR Am J Roentgenol. 2015 Dec;205(6):1288-94. doi: 10.2214/AJR.15.14299. PMID 26587936
- [Background] Fakhry C, Agrawal N, Califano J, Messing B, Liu J, Saunders J, Ha P, Coquia S, Hamper U, Gillison M, Blanco R. The use of ultrasound in the search for the primary site of unknown primary head and neck squamous cell cancers. Oral Oncol. 2014 Jul;50(7):640-5. doi: 10.1016/j.oraloncology.2014.03.015. Epub 2014 May 10. PMID 24819862
- [Background] Kreimer AR, Johansson M, Yanik EL, Katki HA, Check DP, Lang Kuhs KA, Willhauck-Fleckenstein M, Holzinger D, Hildesheim A, Pfeiffer R, Williams C, Freedman ND, Huang WY, Purdue MP, Michel A, Pawlita M, Brennan P, Waterboer T. Kinetics of the Human Papillomavirus Type 16 E6 Antibody Response Prior to Oropharyngeal Cancer. J Natl Cancer Inst. 2017 Aug 1;109(8):djx005. doi: 10.1093/jnci/djx005. PMID 28376197
- [Background] Holzinger D, Wichmann G, Baboci L, Michel A, Hofler D, Wiesenfarth M, Schroeder L, Boscolo-Rizzo P, Herold-Mende C, Dyckhoff G, Boehm A, Del Mistro A, Bosch FX, Dietz A, Pawlita M, Waterboer T. Sensitivity and specificity of antibodies against HPV16 E6 and other early proteins for the detection of HPV16-driven oropharyngeal squamous cell carcinoma. Int J Cancer. 2017 Jun 15;140(12):2748-2757. doi: 10.1002/ijc.30697. Epub 2017 Apr 4. PMID 28316084
- [Background] Lang Kuhs KA, Pawlita M, Gibson SP, Schmitt NC, Trivedi S, Argiris A, Kreimer AR, Ferris RL, Waterboer T. Characterization of human papillomavirus antibodies in individuals with head and neck cancer. Cancer Epidemiol. 2016 Jun;42:46-52. doi: 10.1016/j.canep.2016.03.003. Epub 2016 Mar 21. PMID 27010729